CLINICAL TRIAL: NCT02534974
Title: Impact of the Addition of a Device Providing Continuous Pneumatic Regulation of Tube Cuff Pressure to an Overall Strategy Aimed at Preventing Ventilator-associated Pneumonia in the Severe Trauma Patient. A Multicentre, Randomised, Controlled Study.
Acronym: AGATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: AGATE
Record Dates: First submitted 2015-07-28; First posted 2015-08-28 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2018-04

CONDITIONS: Ventilation-associated Pneumonia; Severe Trauma Patient
Keywords: Critical care; Trauma patients

INTERVENTIONS:
Device: NOSTEN
  Other Names: device providing continuous pneumatic regulation of tube cuff pressure

SUMMARY:
Ventilation-associated pneumonia is the main site of healthcare-associated infections in the severe trauma patient, with a mean incidence rate of 35%. Ventilator-associated pneumonia increases morbi-mortality, length of stay in intensive care and overall management costs. As was recalled by the jury of the 2008 SFAR-SRLF consensus conference on the prevention of nosocomial infections contracted in intensive care, success in this preventive endeavour depends on a number of measures: orotracheal intubation route, maintaining tube cuff pressure between 25 and 30 cm H2O, maintaining a semi-seated position ≥30°, nasal and oropharyngeal care at regular intervals, striving to avoid unscheduled extubation, and use of a written sedation-analgesia algorithm allowing for early weaning from ventilation.

Devices ensuring continuous pneumatic control of tube cuff pressure are more efficient in maintaining tracheal balloon pressure than intermittent adjustments using a hand-held manometer. In one study, these devices clearly facilitated diminution of microaspiration of gastric contents and of ventilator-associated pneumonia incidence density (9.7 vs. 22 VAP/1000 days of mechanical ventilation; p = 0.005).

The investigators are putting forward the hypothesis that by adjoining a device providing continuous pneumatic regulation of tube cuff pressure to an overall strategy aimed at ventilator-associated pneumonia prevention (including semi-recumbent position ≥30°, oro-nasal-pharyngeal care at regular intervals and reduced risk exposure) can decrease VAP incidence by 50% in severely traumatised patients whose condition necessitates mechanical ventilation of an expected duration exceeding 48h.

Ours is the first large-scale study to evaluate the interest of an innovative technology bundle on decrease of ventilator-associated pneumonia incidence in one of the intensive care populations the most at risk, namely severe trauma patients, a population presently benefiting from the other recommended preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a severe trauma as defined by an Injury Severity Score (ISS) >15,
* Aged at least 18 years,
* Intubated for less than 15h,
* Necessitating recourse to mechanical ventilation for an expected period ≥ 48h,
* Participating in a social security scheme or benefiting from such a scheme by means of a third party.

Exclusion Criteria:

* Patient likely to die over the 48h following admission,
* Nasotracheal intubation,
* Patient intubated through a tracheal tube with subglottic secretion drainage
* Intubation carried out 24h or more after the trauma,
* Ventilation with tracheotomy,
* Refusal to participate in the research,
* Contraindication to the head-up position,
* Participation in another research protocol focusing on an anti-infective treatment or on a measure decreasing the risk of infection,
* Persons benefiting from reinforced protection or persons deprived of freedom subsequent to a legal or administrative decision, minors under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having developed VAP at D28 in intensive care according to the ATS definition | 28 days

SECONDARY OUTCOMES:
Proportion of patients having developed VAP in ICU according to the ATS definition | max 60 days
Proportion of patients having developed early (≤ day 7) or late (> day 7) VAP in ICU according to the ATS definition | max 60 days
Time to first episode of VAP diagnosis according to the ATS definition | max 60 days
Proportion of patients developing ventilator-associated events (VAE) according to the CDC definition | max 60 days
Number of ventilator free days | max 60 days
Number of antibiotic free days | max 60 days
ICU length-of-stay | max 60 days
Proportion of patient who died during their ICU stay | max 60 days
Proportion of patients requiring corticosteroids or bronchodilators within 48 hours of tracheal extubation | max 60 days

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Sigismond LASOCKI, Angers
  - Sébastien PILI FLOURY, Besançon
  - Jean Michel CONSTANTIN, Clermont-Ferrand
  - Catherine PAUGAM, Clichy
  - Belaid BOUHEMAD, Dijon
  - Dominique FALCON, Grenoble
  - Marc LEONE, Marseille
  - Karim ASEHNOUNE, Nantes
  - Carole ICHAI, Nice
  - Jean Yves LEFRANT, Nîmes
  - Olivier MIMOZ, Poitiers
  - Benoit VEBER, Rouen
  - Julien POTTECHER, Strasbourg

REFERENCES:
- [Derived] Marjanovic N, Boisson M, Asehnoune K, Foucrier A, Lasocki S, Ichai C, Leone M, Pottecher J, Lefrant JY, Falcon D, Veber B, Chabanne R, Drevet CM, Pili-Floury S, Dahyot-Fizelier C, Kerforne T, Seguin S, de Keizer J, Frasca D, Guenezan J, Mimoz O; AGATE Study Group. Continuous Pneumatic Regulation of Tracheal Cuff Pressure to Decrease Ventilator-associated Pneumonia in Trauma Patients Who Were Mechanically Ventilated: The AGATE Multicenter Randomized Controlled Study. Chest. 2021 Aug;160(2):499-508. doi: 10.1016/j.chest.2021.03.007. Epub 2021 Mar 13. PMID 33727034
- [Derived] Marjanovic N, Frasca D, Asehnoune K, Paugam C, Lasocki S, Ichai C, Lefrant JY, Leone M, Dahyot-Fizelier C, Pottecher J, Falcon D, Veber B, Constantin JM, Seguin S, Guenezan J, Mimoz O; AGATE study group. Multicentre randomised controlled trial to investigate the usefulness of continuous pneumatic regulation of tracheal cuff pressure for reducing ventilator-associated pneumonia in mechanically ventilated severe trauma patients: the AGATE study protocol. BMJ Open. 2017 Aug 7;7(8):e017003. doi: 10.1136/bmjopen-2017-017003. PMID 28790042